CLINICAL TRIAL: NCT03959696
Title: Promoting Informed Decisions About Colorectal Cancer Screening in Older Adults (PRIMED Study): Randomized Trial
Brief Title: Promoting Informed Decisions About Cancer Screening in Older Adults
Acronym: PRIMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: MaineHealth (Other); Brigham and Women's Hospital (Other); Newton-Wellesley Hospital (Other); North Shore Medical Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018P002848; CDR-2017C3-9270 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2019-05-01; First posted 2019-05-22 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Screening
Keywords: Shared Decision Making; Patient Reported Outcomes; Continuing Medical Education; early detection of cancer; colonoscopy; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-arm, multi-site cluster randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Physician participants will not be blinded to the study arm. Patients will not be given any information on their physician's assigned arm. Statistician will be blinded to the assignment when analyzing the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Notification only arm (Active Comparator): Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Interventions: Behavioral: Notification
- Training and Notification arm (Experimental): Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Interventions: Behavioral: Notification; Behavioral: Training

INTERVENTIONS:
Behavioral: Notification — Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
Behavioral: Training — The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
  Arms: Training and Notification arm

SUMMARY:
This project aims to examine the impact of different interventions designed to help individualize colorectal cancer (CRC) screening decisions in adults aged 76-85. Clinicians will be assigned by chance to one of two arms. In the Intervention arm, clinician participants will complete a training course and will also be notified of patients in the target age group who are due for a discussion about CRC screening. In the Comparator arm, clinician participants will be notified of their patients in the target age group with an upcoming visit who are due for a discussion about CRC screening. The investigators expect that patients seen by clinicians in the intervention arm will report more involvement in the decision making process, be more knowledgeable about the risks and benefits of CRC screening, and will have better quality decisions. Further, the investigators expect that the physicians in the intervention arm will have greater confidence in and demonstrate more skills for conducting shared decision making conversations as compared to those in the control arm.

DETAILED DESCRIPTION:
This study will advance understanding of how to engage and inform older adults in decisions about whether to continue or stop colorectal cancer (CRC) screening. The study will randomly assign about 50 primary care clinicians from 5 different sites to one of two different arms. In the Intervention arm, clinician participants will complete a training course and will also be notified of patients aged 76-85 with an upcoming visit who are due for a discussion about CRC screening. In the Comparator arm, clinician participants will be notified of their patients in the target age group with an upcoming visit who are due for a discussion about CRC screening. The study staff will collect surveys from about 500 eligible patients of participating physicians shortly after their visit to determine the impact of the intervention on patient-reported measures including the amount of shared decision making, knowledge, and preferences for cancer screening. Study staff will follow patients to track colorectal cancer screening tests in the 12 months following the visit and will survey some patients again at 12 months to examine any barriers to follow through with their preferred approach. The study will also assess physician's ability to demonstrate shared decision making skills for cancer screening decisions in simulated patient interactions. Caregivers, if identified by a patient participant, will also complete a short survey evaluating the visit.

ELIGIBILITY:
For Clinicians, eligibility will not be decided by sex, gender, or age

Inclusion Criteria for clinicians:

* Primary Care Physician (MD or NP)
* Manages a panel of patients
* Has ≥20 potentially eligible patients (age 76-85 and due for colorectal cancer screening) in their panel
* Practices at participating site

Exclusion Criteria for clinicians:

* Residents, medical students
* Does not manage panel of patients (e.g. urgent care clinician)

Patients of participating clinicians will be enrolled to evaluate the impact of the interventions.

Inclusion Criteria for patients:

* Adults, age 76-85 at the time of the scheduled visit
* Scheduled for non-urgent office visit with a participating clinician during the study period
* Due or overdue for colorectal cancer screening (e.g. never been screened, 1 year or less to follow-up interval indicated on previous test).

Exclusion Criteria for patients:

* Prior diagnosis of colon or rectal cancer, inflammatory bowel disease or genetic disorder that raises CRC risk (e.g. hereditary non-polyposis CRC and familial adenomatous polyposis)
* Unable to consent for themselves (e.g. moderate to severe dementia or other major cognitive limitations)
* Unable to read or write in English or Spanish

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen R Sepucha, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Leigh Simmons, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - North Shore Medical Center, Danvers, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
To promote research replicability, transparency and future use of the data, de-identified data sets of the patient and clinician survey data will be created and will be available, by request, to outside researchers.
  After the main manuscripts have been published, de-identified data sets will also be deposited in an open access service such as, ICPSR (https://www.icpsr.umich.edu/icpsrweb/). Before a dataset is made available for access, ICPSR completes a detailed review of all datasets to assess disclosure risk. If necessary, ICPSR modifies data to reduce disclosure risk or limits access to datasets for which modifying the data would substantially limit their utility or the risk of disclosure remains high. No information that contains identifiers or that could be used to link an individual to the data will be included in the de-identified data set.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Three months after the end of the funded grant period, the study materials and de-identified data will be available, by request, from the PI. Once data are placed on an open access service such as ICPSR they will be available indefinitely.
Access Criteria: The PI will share a de-identified data set with outside investigators at no cost, according to approved Partners and Massachusetts General Hospital policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.
  On ICPSR, individuals must register and agree to ICPSR's Responsible Use statement prior to accessing datasets.

REFERENCES:
- [Derived] Sepucha KR, Chang Y, Valentine KD, Atlas SJ, Han PKJ, Leavitt LJ, Mancini B, Richter JM, Siegel LC, Fairfield KM, Simmons LH. Shared Decision-Making in Colorectal Cancer Screening for Older Adults: A Secondary Analysis of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2429645. doi: 10.1001/jamanetworkopen.2024.29645. PMID 39178001
- [Derived] Sepucha K, Han PKJ, Chang Y, Atlas SJ, Korsen N, Leavitt L, Lee V, Percac-Lima S, Mancini B, Richter J, Scharnetzki E, Siegel LC, Valentine KD, Fairfield KM, Simmons LH. Promoting Informed Decisions About Colorectal Cancer Screening in Older Adults (PRIMED Study): a Physician Cluster Randomized Trial. J Gen Intern Med. 2023 Feb;38(2):406-413. doi: 10.1007/s11606-022-07738-4. Epub 2022 Aug 5. PMID 35931908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May - August 2019, physicians enrolled onto the study from Internal Medicine and Family Medicine practices affiliated with five hospital networks-three academic medical centers and two community hospitals in the Northeast US. We targeted about 10 patients per physician from October 2019-April 2021. We anticipated enrolling 500 patients. Enrolled patients were able to invite a companion, if applicable
Groups:
- Notification Only Arm/Providers: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
- Notification Only Arm/Patients: Eligible patients who completed a visit with a participating physician in the 'notification only' arm.
  Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
- Training and Notification Arm/Providers: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
- Training and Notification Arm/Patients: Eligible patients who completed a visit with a participating physician in the 'training and notification' arm.
  Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
- Notification Only Arm/Companion; Training and Notification Arm/Companion: Enrolled patients were able to invite a companion, if applicable
Period: Overall Study
Arm/Group | Notification Only Arm/Providers | Notification Only Arm/Patients | Training and Notification Arm/Providers | Training and Notification Arm/Patients | Notification Only Arm/Companion | Training and Notification Arm/Companion
Started | 31 | 230 | 28 | 236 | 5 | 6
Completed | 31 | 230 | 28 | 236 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Training and Notification Only Arm/Patients: Eligible patients who completed a visit with a participating physician in the 'training and notification' arm.
  Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
- Notification Only Arm / Companions; Training and Notification Arm/ Companions: Enrolled patients were able to invite a companion, if applicable
- Total: Total of all reporting groups
Arm/Group | Notification Only Arm/Providers | Notification Only Arm/Patients | Training and Notification Arm/Providers | Training and Notification Only Arm/Patients | Notification Only Arm / Companions | Training and Notification Arm/ Companions | Total
Number analyzed (Participants) | 31 | 230 | 28 | 236 | 5 | 6 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The analytic set are the eligible patients who completed a survey. Three patients were removed after determining they did not meet eligibility criteria.
  years | 52.4 (9.0) | 79.2 (2.8) | 53.1 (10.0) | 79.5 (2.8) | 70 (11) | 77 (12) | 79.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The patients who completed a survey
  Participants
    Female | 16 | 111 | 14 | 138 | 4 | 3 | 286
    Male | 15 | 119 | 14 | 98 | 1 | 3 | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analytic subset are the eligible patients who completed a survey. 3 patients were late ineligible due to: other major health issue, up to date on screening, returned survey too late.
  Participants
    Hispanic or Latino | 0 | 2 | 0 | 4 | 0 | 0 | 6
    Not Hispanic or Latino | 30 | 222 | 28 | 229 | 0 | 0 | 509
    Unknown or Not Reported | 1 | 6 | 0 | 3 | 5 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analytic subset are the eligible patients who completed a survey. 3 patients were late ineligible due to: other major health issue, up to date on screening, returned survey too late.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 7 | 1 | 4 | 3 | 0 | 0 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 4 | 0 | 4 | 0 | 0 | 10
    White | 22 | 215 | 24 | 219 | 0 | 0 | 480
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 10 | 0 | 10 | 5 | 6 | 31
Region of Enrollment [Number; unit: participants] — Population: The patients and companions who completed a survey. The physicians who enrolled patients.
  participants
    United States | 31 | 230 | 28 | 236 | 5 | 6 | 536

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Process (SDMP) Scale Score
Description: The SDMP scale is a short, patient-reported scale that asks patients about discussion of options, pros and cons of colonoscopy and discussion of patients' preferences. Total scores range from 0-4, with higher scores indicating more shared decision making.
Time Frame: About 1 week after the physician visit
Population: This analytic sample includes patients who completed the survey and completed data on all four SDM Process questions.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Notification Only Arm/ Patients: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
- Training and Notification Arm/ Patients: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
Arm/Group | Notification Only Arm/ Patients | Training and Notification Arm/ Patients
Number analyzed (Participants) | 222 | 232
Score on a scale | 1.1 (1.2) | 1.5 (1.2)
Statistical Analysis 1: Comparison: Notification Only Arm/ Patients vs Training and Notification Arm/ Patients; The null hypothesis SDMP is equal in the two arms; Test type: Superiority; p = .011, Regression, Linear — A priori threshold for statistical significance is .05; We used a linear regression model with Generalized Estimating Equations (GEE) techniques to account for the patients-within-physicians data structure; Mean Difference (Net) = .36, 95% CI 2-sided [.08 to .64] — Mean difference is the Training + Notification arm minus the Notification only arm

2. Secondary Outcome: Patients' Colorectal Cancer Screening Knowledge Score
Description: Colorectal Cancer (CRC) Screening Knowledge will be assessed with multiple choice knowledge items adapted from the CRC Decision Quality Instrument. A total score from 0-100% will be calculated based on the number of correct answers, with higher scores indicating higher knowledge.
Time Frame: 1 week after physician visit
Population: The data is of patients who answered at least 4 of the 7 questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Notification Only Arm/ Patients | Training and Notification Arm/ Patients
Number analyzed (Participants) | 221 | 228
score on a scale | 61 (18.8) | 63 (17.7)
Statistical Analysis 1: Comparison: Notification Only Arm/ Patients vs Training and Notification Arm/ Patients; The null hypothesis is that the two arms have the same knowledge score; Test type: Superiority; p = 0.36, Regression, Linear — A priori threshold for statistical significance is .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.77, 95% CI 2-sided [-2.01 to 5.55]

3. Secondary Outcome: Percentage of Patients Who Received Preferred Approach to Colorectal Cancer Testing
Description: Colorectal Cancer Screening Preference assessed with 1 item adapted from the CRC Decision Quality Instrument will be compared with the screening approach followed (assessed via chart review and patient report) to determine the percentage of patients who received preferred approach to testing.
Time Frame: 1 week after physician visit (preference); 12 months after physician visit (testing)
Population: 450 patients who indicated a clear preference on the post visit survey were analyzed. The population excludes 4 who indicated 'other' and 12 who did not answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Notification Only Arm/ Patients | Training and Notification Arm/ Patients
Number analyzed (Participants) | 223 | 227
Participants | 103 | 115
Statistical Analysis 1: Comparison: Notification Only Arm/ Patients vs Training and Notification Arm/ Patients; We will compare the percentages of patients who received their preferred screening in the 12 months after the visit across the two groups using logistic regression model with the GEE approach to adjust for clustering of patients within clinicians; Test type: Superiority — We will have 81% power to detect a difference of 14% in rates (e.g. decrease from 61% to 47%); p = 0.47, Regression, Logistic

4. Secondary Outcome: Physician's Shared Decision Making Skills
Description: The transcripts from the simulated patient interactions will be scored by two coders using Braddock's Informed Decision Making framework. Total scores range from 0-9 with higher scores indicating more shared decision making elements in the interaction.
Time Frame: Baseline
Population: Physicians who completed a recorded simulated patient interaction with a standardized patient.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Training and Notification Arm/ Providers: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
Arm/Group | Notification Only Arm/Providers | Training and Notification Arm/ Providers
Number analyzed (Participants) | 26 | 28
Score on a scale | 5.5 (1.3) | 6.1 (1.6)
Statistical Analysis 1: Comparison: Notification Only Arm/Providers vs Training and Notification Arm/ Providers; Test type: Superiority; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = 0.53

5. Secondary Outcome: Colorectal Cancer Screening Rates
Description: The chart review results of cancer screening rates for patients enrolled in the study.
Time Frame: 1 year
Population: 466 enrolled patients whose chart was reviewed for completion of cancer screening
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Notification Only Arm/Patients: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
- Training and Notification Arm/Patients: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
Arm/Group | Notification Only Arm/Patients | Training and Notification Arm/Patients
Number analyzed (Participants) | 230 | 236
percentage of participants | 29.1 [23.3 to 35.5] | 38.6 [32.3 to 45.1]
Statistical Analysis 1: Comparison: Notification Only Arm/Patients vs Training and Notification Arm/Patients; Null hypothesis was equal screening rate in both arms; Test type: Superiority; p = 0.032, Chi-squared; Risk Difference (RD) = 9.4, 95% CI 2-sided [0.9 to 18.0]

6. Secondary Outcome: Clinician Satisfaction With the Visit
Description: The percentage of study patient visits where the clinicians' reported that they were 'extremely or very satisfied' will be compared across arms.
Time Frame: 1 week post visit
Population: 59 participating physicians completed post-visit surveys for 376 participating patients.
Measure: Count of Participants; unit: Participants
Groups:
- Notification Only Arm/Patient: Eligible patients who completed a visit with a participating physician in the 'notification only' arm.
  Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
- Training and Notification Arm/Patient: Eligible patients who completed a visit with a participating physician in the 'training and notification' arm.
  Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
Arm/Group | Notification Only Arm/Patient | Training and Notification Arm/Patient
Number analyzed (Participants) | 176 | 200
Participants | 138 | 171
Statistical Analysis 1: Comparison: Notification Only Arm/Patient vs Training and Notification Arm/Patient; Test type: Superiority; p = 0.64, Chi-squared; Risk Difference (RD) = 1.5

7. Other Pre Specified Outcome: Companion SDM Process Scale Score
Description: Companions will complete an adapted version of the SDM Process survey to provide a different perspective on the conversation and involvement of the patient. A total score will range from 0-4, with higher scores indicating more shared decision making.
Time Frame: About a week after physician visit
Population: Very few patients indicated that they had a companion (spouse, friend, family member) with them at the visit. If a name was provided, companions were contacted and ask to complete a post-visit survey. 11 companions were identified, but only 10 completed the SDM Process questions.
Measure: Mean (Standard Deviation); unit: Score on a scale of 0-4
Groups:
- Notification Only Arm/Companion: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
- Training and Notification Arm/Companion: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening and will complete a two-hour shared decision making communication skills training course that includes case studies, interactive exercises, and lecture content.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
  Training: The 2-hour continuing medical education course in shared decision making, simulated patient interaction to practice skills, and monthly calls for a year to review difficult cases with clinical and shared decision making experts.
Arm/Group | Notification Only Arm/Companion | Training and Notification Arm/Companion
Number analyzed (Participants) | 5 | 6
Score on a scale of 0-4 | 2.1 (1.3) | 1.9 (1.2)

8. Other Pre Specified Outcome: Clinician Attitude Toward Shared Decision Making
Description: The investigators will use five items to assess clinicians' confidence in Shared Decision Making Skills and Barriers to SDM. A total confidence score (0-20) with higher scores indicating higher confidence and a barrier score (0-8) higher scores indicating more barriers will be calculated.
Time Frame: Baseline
Population: Comparator physicians' reported confidence of shared decision making and barriers to shared decision making on a baseline survey is compared to Intervention physicians' reported confidence of shared decision making and barriers to shared decision making after completion of the training webinar.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Notification Only Arm/Providers | Training and Notification Arm/ Providers
Number analyzed (Participants) | 33 | 34
Score on a scale
  Total Confidence | 10.2 (2.4) | 10.7 (1.8)
  Barrier Confidence | 0.79 (1.4) | 0.88 (1.57)

ADVERSE EVENTS:
Time Frame: patients were followed for 1 year
Groups:
- Notification Only/Providers: Clinician participants will be notified of their patients aged 76-85 with an upcoming visit who are due for colorectal cancer screening.
  Notification: Clinicians will be notified of their patients aged 76-85 with an upcoming, non urgent visit who are due for colorectal cancer screening.
- Training and Notification Arm/Companions; Notification Only/Companions: Enrolled patients were able to invite a companion, if applicable
Arm/Group | Notification Only/Providers | Notification Only Arm/Patients | Training and Notification Arm/Providers | Training and Notification Arm/Patients | Training and Notification Arm/Companions | Notification Only/Companions
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/230 | 0/28 | 0/236 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/230 | 0/28 | 0/236 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/31 | 0/230 | 0/28 | 0/236 | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03959696/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03959696/SAP_001.pdf